CLINICAL TRIAL: NCT03682601
Title: Sinecatechins Ointment, a Botanical Drug Derived From Green Tea, for the Treatment of Significant to Severe Secondary Provoked Vestibulodynia in Sexually Active, Post-Menopausal Women With Vulvovaginal Atrophy
Brief Title: Sexual Penetration Pain in Postmenopausal Women: A Topical Botanical Drug Treatment
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: pandemic
Sponsor: GTO Pharmaceutical, LLC (Other)
Responsible Party: Principal Investigator, Lila Nachtigall, M.D., Lila Nachtigall, M.D., Professor of Gynecology, Dr. Lila Nachtigall Rapid Medical Research, New York
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GTO1
Record Dates: First submitted 2018-09-14; First posted 2018-09-24 (Actual); Results first posted 2022-06-28 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Sexual Pain Disorders; Postmenopausal Symptoms; Vulvovaginal Atrophy; Female Sexual Dysfunction; Dyspareunia; Vulvodynia; Vestibulodynia; Arousal Disorders, Sexual; Genito-Pelvic Pain/Penetration Disorder; Female Sexual Arousal Disorder
Keywords: Sexual Pain; Postmenopausal Symptoms; Vulvovaginal Atrophy; Vulvodynia; Dyspareunia; Vestibulodynia; Female Sexual Dysfunction; Arousal Disorders, Sexual; Painful Penetration; Painful intercourse; Vulvar Pain; Pain at vaginal opening; Entrance Pain; Lack of Lubrication; Lack of Arousal
MeSH Terms: conditions — Dyspareunia; Vulvodynia; Sexual Dysfunctions, Psychological | interventions — polyphenon E; Petrolatum

STUDY DESIGN:
Intervention Model Description: Randomized, Double Blinded, Placebo Controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Placebo (Placebo Comparator): 15 postmenopausal women will apply a 1/2 inch strand of Placebo ointment once daily to their vulvar vestibule for a total of 4 weeks.
  They will come for three office visits with the gynecologist, who will exam their vulvar vestibule and perform a Qtip test. The Qtip test consists of applying pressure with a cotton tipped swab to the vulvar vestibule and asking the participant to rate the degree of pain that they experience on a scale from 0-10 ( 0=no pain; 1-3=mild pain; 4-6=moderate pain; 7-9=significant pain; 10=severe pain).
  A swab will be taken of the lateral vaginal wall for to assess the degree of vaginal atrophy.
  The participant will fill out questionnaire during office visits with the gynecologist. In addition, questionnaire will be filled out online on a HIPAA compliant web based survey at the end of weeks 1 and 3 and one week after stopping study ointment.
  Interventions: Drug: Placebo
- 5% Topical sinecatechins ointment (Active Comparator): 15 postmenopausal women will apply a 1/2 inch strand of 5% sinecatechins topical ointment once daily to their vulvar vestibule for a total of 4 weeks.
  They will come for three office visits with the gynecologist, who will exam their vulvar vestibule and perform a Qtip test. The Qtip test consists of applying pressure with a cotton tipped swab to the vulvar vestibule and asking the participant to rate the degree of pain that they experience on a scale from 0-10 ( 0=no pain; 1-3=mild pain; 4-6=moderate pain; 7-9=significant pain; 10=severe pain).
  A swab will be taken of the lateral vaginal wall for to assess the degree of vaginal atrophy.
  The participant will fill out questionnaire during office visits with the gynecologist. In addition, questionnaire will be filled out online on a HIPAA compliant web based survey at the end of weeks 1 and 3 and one week after stopping study ointment.
  Interventions: Drug: 5% sinecatechins ointment
- 10% Topical sinecatechins ointment (Active Comparator): 15 postmenopausal women will apply a 1/2 inch strand of 10% sinecatechins topical ointment once daily to their vulvar vestibule for a total of 4 weeks.
  They will come for three office visits with the gynecologist, who will exam their vulvar vestibule and perform a Qtip test. The Qtip test consists of applying pressure with a cotton tipped swab to the vulvar vestibule and asking the participant to rate the degree of pain that they experience on a scale from 0-10 ( 0=no pain; 1-3=mild pain; 4-6=moderate pain; 7-9=significant pain; 10=severe pain).
  A swab will be taken of the lateral vaginal wall for to assess the degree of vaginal atrophy.
  The participant will fill out questionnaire during office visits with the gynecologist. In addition, questionnaire will be filled out online on a HIPAA compliant web based survey at the end of weeks 1 and 3 and one week after stopping study ointment.
  Interventions: Drug: 10% sinecatechins ointment

INTERVENTIONS:
Drug: 5% sinecatechins ointment — Topical 5% sinecatechins ointment will be applied once daily.
  Other Names: Veregen ointment
  Arms: 5% Topical sinecatechins ointment
Drug: Placebo — Aquaphor/vehicle
  Other Names: Aquaphor
  Arms: Placebo
Drug: 10% sinecatechins ointment — Topical 10% sinecatechins ointment will be applied three times per week up to once daily.
  Other Names: Veregen ointment
  Arms: 10% Topical sinecatechins ointment

SUMMARY:
This study will evaluate the use of topical 5 or 10% sinecatechins, a botanical drug derived from green tea for the alleviation of sexual pain in the area around the vaginal opening (the vulvar vestibule), that is a main source of pain during sexual contact or dyspareunia, in postmenopausal women, with vulvovaginal atrophy. Women may or may not be using estrogens. Half of the women will receive the study drug, 5 or 10% sinecatechins and half will receive placebo. In addition to the reduction or elimination of pain upon penetration, women may also experience increase in lubrication, arousal and intensity of orgasm

DETAILED DESCRIPTION:
Topical Veregen (15% sinecatechins) is an FDA approved botanical drug derived from green tea and is approved to be used as multiple doses, three times a day to treat all visible external genital warts.

Topical green tea ointment has been shown to alleviate pain and improve wound healing in the vulvar vestibule for women who have had a recent episiotomy in the medical literature. In private clinical practice, dilute Veregen, sinecatechins ointment, has been effective in alleviating , sexual pain, vulvar vestibular pain, dyspareunia, in postmenopausal women as well as improving overall sexual satisfaction,( increasing lubrication, arousal and quality of orgasm). In this study, dilute Veregen, (5 or 10% sinecatechins) or placebo is being applied, as a single dose, topically, three times/week up to once a day, to alleviate pain in the vulvar vestibule, penetration pain, upon sexual contact or other manipulation of this area in postmenopausal women. Women are eligible whether or not they are currently using any form of estrogen or other hormonal treatments (eg. DHEA). Please note that women not using estrogen or who maybe taking aromatase inhibitors, tamoxifen, SERMS, are also eligible to be included.

ELIGIBILITY:
Inclusion Criteria:

Generally healthy women must meet the following eligibility criteria:

1. For surgically menopausal women, be 20-70 years of age and at least 12 months post menopause.
2. For naturally postmenopausal women, be 40-70 years of age and at least 1 year post menopause (defined as no spontaneous menses for 1 year).
3. Women taking estrogens may enroll in the trial.
4. For women who are not taking any estrogen or who are taking an aromatase inhibitor, In screening their vaginal power of hydrogen (pH) will be 4.6 or greater and their vaginal maturation index will be consistent with vaginal atrophy. Vaginal atrophy is thinning, drying and of the vaginal walls due to having less estrogen in the body.
5. Be, sexually functional, both psychologically and physically, whereby a woman is to be psychologically interested in sexual activity and (unless these activities are precluded by pain) is physically sexually active with regular vestibular including vaginal introital genital manipulation whether through masturbation or partner sex, whether using digits, oral sexual contact, sex toys, and/or penile penetration present at regular intervals each month during the 4-week pre-treatment and the 4- week active treatment period of the study and ending at the 6th- week of their participation in the study.
6. Be able and willing to participate in the study as evidenced by providing written informed consent.
7. Answer affirmatively to all of the following questions:

   1. Before your vulvar pain, would you say that in general, your sex life was good and satisfying?
   2. Since you have been experiencing vulvar pain, do you feel you have experienced a meaningful loss in your desire for sex?
   3. Since experiencing vulvar pain, do you feel you have experienced a significant decrease in your sexual activity?
   4. Are you concerned or bothered by your current level of desire for or interest in sex?
   5. Would you like to see an increase in your level of interest or desire for sex and sexual activity?
8. Women can enter the trial if they are taking estrogens.
9. Women can enter the trial if they are taking DHEA.
10. Women can enter the trial if they are not taking estrogens.
11. Women can enter the trial if they are taking aromatase inhibitors.

Exclusion Criteria:

1. Have any physical limitations or sexual trauma that would interfere with normal sexual function.
2. Have used within the last 12 weeks any of the following medications/preparations that may interfere with the study purpose: systemic corticosteroids (acute use for fewer than 7 days is accepted), SSRI's, tricyclic antidepressants, anti-androgens, spironolactone, phosphodiesterase type 5 (PDE5) inhibitors (Viagra ®).
3. Be experiencing any chronic or acute life stress relating to any major life change, such as recent loss of income or the death of a close family member, that may, in the opinion of the Investigator, significantly interfere with sexual function.
4. Have significant psychiatric disorder, a significant alcohol or drug dependency and/or be receiving pharmacologic treatment for such illness or disorder.
5. Have evidence of clinically significant organic disorder on the history and/or physical examination that would, in the opinion of the Investigator, put the patient at risk, present the patient from completing the study, or otherwise affect the outcome of the study.
6. Have a history of genital herpes because of the episodic nature of genital herpes and of the known possibility of occurrence of herpetic pain without visible dermatologic manifestations of herpes. Genital herpes and its accompanying genital pain may obscure the source of the genital pain experienced and confound the ability to determine the efficacy of treatment/placebo on endpoint of alleviation of pain in women with secondary provoked vulvar vestibular pain.
7. Have any infection of the genitalia
8. Have lichen sclerosis, lichen planus, contact dermatitis, psoriasis or any inflammatory condition or abrasions of the vulva
9. Have an episiotomy scar in the area where pain is perceived as it may confound the etiology of the perceived pain
10. Have diabetes.

    -

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Participant must be a postmenopausal female who has not menstruated for at least one year either because of surgical removal of ovaries and uterus or because of natural menopause. Women taking estrogens, DHEA, can continue to use them during the clinical trial. Women not taking estrogens or are on aromatase inhibitors can enter the trial.
Enrollment: 32 (Actual)
Dates: Start 2018-08-30 (Actual); Primary Completion 2021-02-12 (Actual); Study Completion 2021-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lila Nachtigall, M.D., Principal Investigator — Rapid Medical Research, New York
Locations (4):
- United States (4):
  - Lila Nachtigall, M.D., New York, New York
  - Miriam Greene, M.D., New York, New York
  - Cynthia Krause, M.D., New York, New York
  - Janis Enzenbacher, M.D., Nyack, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shahrahmani H, Kariman N, Jannesari S, Rafieian-Kopaei M, Mirzaei M, Ghalandari S, Shahrahmani N, Mardani G. The effect of green tea ointment on episiotomy pain and wound healing in primiparous women: A randomized, double-blind, placebo-controlled clinical trial. Phytother Res. 2018 Mar;32(3):522-530. doi: 10.1002/ptr.5999. Epub 2017 Dec 13. PMID 29235159
- [Background] Goetsch MF, Lim JY, Caughey AB. Locating pain in breast cancer survivors experiencing dyspareunia: a randomized controlled trial. Obstet Gynecol. 2014 Jun;123(6):1231-1236. doi: 10.1097/AOG.0000000000000283. PMID 24807329

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: 15 postmenopausal women will apply a 1/2 inch strand of Placebo ointment once daily to their vulvar vestibule for a total of 4 weeks.
  They will come for three office visits with the gynecologist, who will exam their vulvar vestibule and perform a Qtip test. The Qtip test consists of applying pressure with a cotton tipped swab to the vulvar vestibule and asking the participant to rate the degree of pain that they experience on a scale from 0-10 ( 0=no pain; 1-3=mild pain; 4-6=moderate pain; 7-9=significant pain; 10=severe pain).
  A swab will be taken of the lateral vaginal wall for to assess the degree of vaginal atrophy.
  The participant will fill out questionnaire during office visits with the gynecologist. In addition, questionnaire will be filled out online on a HIPAA compliant web based survey at the end of weeks 1 and 3 and one week after stopping study ointment.
  Placebo: Aquaphor/vehicle
- 5% Topical Sinecatechins Ointment: 15 postmenopausal women will apply a 1/2 inch strand of 5% sinecatechins topical ointment once daily to their vulvar vestibule for a total of 4 weeks.
  They will come for three office visits with the gynecologist, who will exam their vulvar vestibule and perform a Qtip test. The Qtip test consists of applying pressure with a cotton tipped swab to the vulvar vestibule and asking the participant to rate the degree of pain that they experience on a scale from 0-10 ( 0=no pain; 1-3=mild pain; 4-6=moderate pain; 7-9=significant pain; 10=severe pain).
  A swab will be taken of the lateral vaginal wall for to assess the degree of vaginal atrophy.
  The participant will fill out questionnaire during office visits with the gynecologist. In addition, questionnaire will be filled out online on a HIPAA compliant web based survey at the end of weeks 1 and 3 and one week after stopping study ointment.
  5% sinecatechins ointment: Topical 5% sinecatechins ointment will be applied once daily.
- 10% Topical Sinecatechins Ointment: 15 postmenopausal women will apply a 1/2 inch strand of 10% sinecatechins topical ointment once daily to their vulvar vestibule for a total of 4 weeks.
  They will come for three office visits with the gynecologist, who will exam their vulvar vestibule and perform a Qtip test. The Qtip test consists of applying pressure with a cotton tipped swab to the vulvar vestibule and asking the participant to rate the degree of pain that they experience on a scale from 0-10 ( 0=no pain; 1-3=mild pain; 4-6=moderate pain; 7-9=significant pain; 10=severe pain).
  A swab will be taken of the lateral vaginal wall for to assess the degree of vaginal atrophy.
  The participant will fill out questionnaire during office visits with the gynecologist. In addition, questionnaire will be filled out online on a HIPAA compliant web based survey at the end of weeks 1 and 3 and one week after stopping study ointment.
  10% sinecatechins ointment: Topical 10% sinecatechins ointment will be applied three times per week up to once daily.
Period: Overall Study
Arm/Group | Placebo | 5% Topical Sinecatechins Ointment | 10% Topical Sinecatechins Ointment
Started | 12 | 7 | 13
Completed | 12 | 7 | 13
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 5% Topical Sinecatechins Ointment | 10% Topical Sinecatechins Ointment | Total
Number analyzed (Participants) | 12 | 7 | 13 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 6 | 11 | 27
  >=65 years | 2 | 1 | 2 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 7 | 13 | 32
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White Non-Hispanic | 12 | 7 | 13 | 32
  Black or African American | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Hispanic or Latino | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 7 | 13 | 32
Numerical Rating Scale [Mean (Standard Deviation); unit: units on a scale from 0 to 10] — Scale Title: Numerical Pain Scale to measure overall pain perceived from vulvar vestibule.
  Minimum value of scale: 0; Maximum value of scale: 10. Subjects were asked to rate from 0 to 10 pain perceived from their vulvar vestibule.
  The mean (standard deviation) for Numerical Pain Scale at each visit was calculated. A higher Numerical Rating Score means worse outcome and lower Numerical Rating Score means a better outcome. The following Numerical Rating Scale categories for Pain definition were utilized: 0=no pain, 1-3=mild pain, 4-6=moderate pain; 7-9=significant pain and 10=severe pain.
  units on a scale from 0 to 10 | 8.6 (0.9) | 7.6 (1.4) | 8.3 (0.8) | 8.2 (1.0)

OUTCOME MEASURES:

1. Primary Outcome: Numerical Rating Scale for Pain
Description: Scale Title: Numerical Pain Scale to measure overall pain perceived from vulvar vestibule.
  Minimum value of scale: 0; Maximum value of scale: 10. Subjects were asked to rate from 0 to 10 pain perceived from their vulvar vestibule.
  The mean (standard error) for Numerical Pain Scale at each visit was calculated. A higher Numerical Rating Score means worse outcome and lower Numerical Rating Score means a better outcome. The following Numerical Rating Scale categories for Pain definition were utilized: 0=no pain, 1-3=mild pain, 4-6=moderate pain; 7-9=significant pain and 10=severe pain.
Time Frame: Numerical Rating Scale for pain was assessed at Visit 1 (initial visit); Visit 2 (at 2 weeks), and Visit 3 (at 4 weeks).
Measure: Mean (Standard Error); unit: score on a scale from 0 to 10.
Arm/Group | Placebo | 5% Topical Sinecatechins Ointment | 10% Topical Sinecatechins Ointment
Number analyzed (Participants) | 12 | 7 | 13
score on a scale from 0 to 10.
  Visit 1 Numerical Rating Scale for pain | 8.6 (0.3) | 7.6 (0.5) | 8.3 (0.2)
  Visit 2 Numerical Rating Scale for pain | 6.4 (0.6) | 4.0 (0.8) | 6.3 (0.6)
  Visit 3 Numerical Rating Scale for pain | 5.9 (0.6) | 2.4 (0.9) | 2.1 (0.4)

2. Secondary Outcome: Q-tip Test Test for Pain on the Vulvar Vestibule
Description: Scale Title: Q-tip test of vulvar vestibular pain. Minimum value of scale: 0; Maximum value of scale: 10. Subjects were asked to rate from 0 to 10 pain perceived from their vulvar vestibule.
  The mean (standard error) for Q-tip test at each visit was calculated. A higher Q-tip score means worse outcome and lower Numerical Rating Score means a better outcome. The following Q-tip test categories for Pain definition were utilized: 0=no pain, 1-3=mild pain, 4-6=moderate pain; 7-9=significant pain and 10=severe pain.
Time Frame: Q-tip test score for pain was assessed at Visit 1 (initial visit); Visit 2 (at 2 weeks), and Visit 3 (at 4 weeks).
Measure: Mean (Standard Error); unit: score on a scale from 0 to 10.
Groups:
- Placebo: 12 postmenopausal women will apply a 1/2 inch strand of Placebo ointment once daily to their vulvar vestibule for a total of 4 weeks.
  They will come for three office visits with the gynecologist, who will exam their vulvar vestibule and perform a Qtip test. The Qtip test consists of applying pressure with a cotton tipped swab to the vulvar vestibule and asking the participant to rate the degree of pain that they experience on a scale from 0-10 ( 0=no pain; 1-3=mild pain; 4-6=moderate pain; 7-9=significant pain; 10=severe pain).
  A swab will be taken of the lateral vaginal wall for to assess the degree of vaginal atrophy.
  The participant will fill out questionnaire during office visits with the gynecologist. In addition, questionnaire will be filled out online on a HIPAA compliant web based survey at the end of weeks 1 and 3 and one week after stopping study ointment.
  Placebo: Aquaphor/vehicle
- 5% Topical Sinecatechins Ointment: 7 postmenopausal women will apply a 1/2 inch strand of 5% sinecatechins topical ointment once daily to their vulvar vestibule for a total of 4 weeks.
  They will come for three office visits with the gynecologist, who will exam their vulvar vestibule and perform a Qtip test. The Qtip test consists of applying pressure with a cotton tipped swab to the vulvar vestibule and asking the participant to rate the degree of pain that they experience on a scale from 0-10 ( 0=no pain; 1-3=mild pain; 4-6=moderate pain; 7-9=significant pain; 10=severe pain).
  A swab will be taken of the lateral vaginal wall for to assess the degree of vaginal atrophy.
  The participant will fill out questionnaire during office visits with the gynecologist. In addition, questionnaire will be filled out online on a HIPAA compliant web based survey at the end of weeks 1 and 3 and one week after stopping study ointment.
  5% sinecatechins ointment: Topical 5% sinecatechins ointment will be applied once daily.
- 10% Topical Sinecatechins Ointment: 13 postmenopausal women will apply a 1/2 inch strand of 10% sinecatechins topical ointment once daily to their vulvar vestibule for a total of 4 weeks.
  They will come for three office visits with the gynecologist, who will exam their vulvar vestibule and perform a Qtip test. The Qtip test consists of applying pressure with a cotton tipped swab to the vulvar vestibule and asking the participant to rate the degree of pain that they experience on a scale from 0-10 ( 0=no pain; 1-3=mild pain; 4-6=moderate pain; 7-9=significant pain; 10=severe pain).
  A swab will be taken of the lateral vaginal wall for to assess the degree of vaginal atrophy.
  The participant will fill out questionnaire during office visits with the gynecologist. In addition, questionnaire will be filled out online on a HIPAA compliant web based survey at the end of weeks 1 and 3 and one week after stopping study ointment.
  10% sinecatechins ointment: Topical 10% sinecatechins ointment will be applied three times per week up to once daily.
Arm/Group | Placebo | 5% Topical Sinecatechins Ointment | 10% Topical Sinecatechins Ointment
Number analyzed (Participants) | 12 | 7 | 13
score on a scale from 0 to 10.
  Visit 1 Q-tip test score | 7.8 (0.5) | 8.2 (0.5) | 7.7 (0.2)
  Visit 2 Q-tip test score | 6.0 (0.5) | 4.8 (0.8) | 5.8 (0.6)
  Visit 3 Q-tip test score | 5.1 (0.6) | 2.9 (0.8) | 1.9 (0.6)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Placebo | 5% Topical Sinecatechins Ointment | 10% Topical Sinecatechins Ointment
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/7 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/7 | 0/13
Other Adverse Events (participants affected / at risk) | 0/12 | 0/7 | 4/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=12) | 5% Topical Sinecatechins Ointment (N=7) | 10% Topical Sinecatechins Ointment (N=13)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 4 (4) — Four patients reported pruritus and itching with daily application of topical 10% ointment at visit 2 that resolved by visit 3.

LIMITATIONS AND CAVEATS:
Early termination due to Coronavirus disease (COVID-19) pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-13): https://cdn.clinicaltrials.gov/large-docs/01/NCT03682601/Prot_SAP_005.pdf